CLINICAL TRIAL: NCT00005012
Title: Antiviral Activity and Tolerability of PEG-Intron in HIV-Infected Subjects Failing HAART
Brief Title: Safety and Effectiveness of PEG-Intron in HIV-Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Schering-Plough (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: B010; P00737
Record Dates: First submitted 2000-03-29; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-08

CONDITIONS: HIV Infections
Keywords: Interferon Alfa-2b; Lymphocyte Transformation; CD4 Lymphocyte Count; RNA, Viral; Virus Inhibitors; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections | interventions — peginterferon alfa-2b

INTERVENTIONS:
Drug: Peginterferon alfa-2b

SUMMARY:
The purpose of this study is to see if it is effective to give PEG-Intron (PEG-IFN) to HIV-infected patients who are not doing well with their current anti-HIV drug combination (HAART).

DETAILED DESCRIPTION:
At entry, patients undergo HIV genotypic/phenotypic analysis. Patients continue their current antiretroviral regimen but are randomized to receive one of four doses of PEG-IFN or PEG-IFN placebo administered subcutaneously once per week until results of HIV genotyping/phenotyping are available (approximately 4 weeks). Patients who respond with a 0.5 log or greater decrease in HIV RNA at Week 4 have optimized HAART added to their ongoing PEG-IFN regimen and are followed for 24 weeks in an observational study.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Have HIV levels of more than 2000 copies/ml.
* Have failed their current HAART (had a significant increase in their HIV levels with HAART).
* Have a CD4 cell count greater than 200 cells/microL.
* Have had more than 6 months of HAART.
* Have been on their current HAART for at least 6 weeks.
* Agree to use an effective method of birth control during the study.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have a history of a serious mental disorder.
* Are allergic to interferons.
* Are pregnant or breast-feeding.
* Are taking certain medications such as ribavirin, hydroxyurea, and ganciclovir.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250
Dates: Start 2000-03; Study Completion 2000-09

CONTACTS AND LOCATIONS:
Locations (22):
- United States (21):
  - East Bay AIDS Ctr, Berkeley, California
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Dupont Circle Physicians Group, Washington D.C., District of Columbia
  - IDC Research Initiative, Altamonte Springs, Florida
  - Duval County Health Department, Jacksonville, Florida
  - Univ of Miami School of Medicine, Miami, Florida
  - Infectious Diseases Associates, Sarasota, Florida
  - Piedmont Physicians at Vinings, Atlanta, Georgia
  - TRIAD Health Practice, Chicago, Illinois
  - Univ of Maryland Institute of Human Virology, Baltimore, Maryland
  - New England Med Ctr / Div of Geo Med & Infect Disease, Boston, Massachusetts
  - Regions Hosp, Saint Paul, Minnesota
  - Washington Univ, St Louis, Missouri
  - Southwestern New Jersey AIDS Clinical Trials, Camden, New Jersey
  - East Orange Veterans Administration Med Ctr, East Orange, New Jersey
  - Beth Israel Med Ctr, New York, New York
  - Univ Hosps of Cleveland, Cleveland, Ohio
  - MCP Hahnemann Univ, Philadelphia, Pennsylvania
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - Amelia Ct Clinic, Dallas, Texas
  - Joseph C Gathe, Houston, Texas
- San Juan VAMC, San Juan, Puerto Rico